CLINICAL TRIAL: NCT04662476
Title: Effect of Vitamin D Supplementation on Sickle Cell Disease Hospitalisation and Related Complications Among Children in Mulago Hospital: A Randomised Clinical Trial
Brief Title: Vitamin D Supplementation in Children With Sickle Cell Disease
Acronym: VIDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Makerere University (Other)
Responsible Party: Principal Investigator, College of Health Sciences, Professor, Makerere University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-117
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Children With Sickle Cell Disease at Mulago Hospital
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: 331 children will be randomised to the intervention and another 331 to the placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The sachets containing vitamin D will be exactly similar to the ones containing the placebo. Both the intervention and placebo granules will be identical in colour, odour, taste and amount. Children will be randomized into treatment groups by order of entry in the study, based on a pre-determined blinded randomization list created and managed by an independent statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D supplement (Active Comparator): 331 children will each received 60,000IU of vitamin D once a month for 3 months.
  Interventions: Dietary Supplement: Vitamin D3
- Intervention (Active Comparator): The intervention arm will receive vitamin D3.
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D3 supplement

SUMMARY:
Children aged 6 months to 12 years of age will be randomised to receive vitamin D 60,000IU once a month for 3 months or a placebo. The vitamin D will be in form of granules supplied in sachets. The primary study outcomes will be incidence of hospitalisation and change in vitamin D levels following supplementation. Secondary outcomes will include incidence of vaso-occlusive crisis (VOC), acute severe respiratory illness, Vitamin D related Severe adverse events and requirements for blood transfusion

DETAILED DESCRIPTION:
BACKGROUND: More than 75% of all children with sickle cell anemia (SCA) are born in sub-Saharan Africa annually. The hallmark of SCA is haemolytic anaemia and or pain crisis that often require hospitalisation. Interventions to reduce the complications, which are prerequisites for frequent hospitalisations, are needed urgently. Vitamin D deficiency is common in children with SCA and is associated with recurrent vaso-occlusive crisis, blood transfusion, hospitalisation and infections. Routine vitamin D supplementation is not practiced in the care of sickle cell disease patients yet it has been associated with improved bone health and bone mineral density, reduced chronic pain and improved quality of life.

HYPOTHESIS: Vitamin D supplementation will lead to a lower incidence of hospitalisation than placebo in Ugandan children with SCA.

METHODS: The study will be a randomized, placebo-controlled, double blind clinical trial in which 331 Ugandan children with SCA aged 6 months to 12 years inclusive will receive vitamin D (60,000IU granules monthly) and another 331 a placebo (identical to vitaminD in appearance) for 3 months. The primary study outcome will be incidence of hospitalisation. Secondary outcomes will include incidence of vaso-occlusive crisis (VOC), acute severe respiratory illness, Vitamin D related Severe adverse events and requirements for blood transfusion IMPACT: If this trial shows a reduction in hospitalisation, it will be the basis for a multi-site pre-post intervention clinical trial to assess real-world safety and efficacy of Vitamin D in African children with SCA. The monthly administration is easy, and since vitamin D is inexpensive, this trial has the potential to improve the health of hundreds/ thousands of African children with SCA through reduction of infection-related morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Documented sickle cell disease (HbSS supported by hemoglobin electrophoresis results) attending Mulago Hospital Sickle Cell Clinic)
2. Age range of 6 months to 12 years, inclusive, at the time of enrolment
3. Weight at least 5.0 kg at the time of enrolment
4. Willingness to comply with all study-related treatments, evaluations, and follow-up

Exclusion Criteria:

1. Known other chronic medical condition (e.g., HIV, malignancy, Renal & liver disease, active clinical tuberculosis)
2. Severe acute malnutrition determined by impaired growth parameters as defined by WHO weight for length/height less than -3SD.
3. Evidence of Vitamin D supplementation in the past one month (by prescription or drug sample)

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 662 (Estimated)
Dates: Start 2021-05-17 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of hospitalisation among children with SCD supplemented with vitamin D versus placebo. | 3 months follow up
  Number of children hospitalised during the follow up period and number of hospitalisations per child
Effect of vitamin supplementation on serum levels of 25 Hydroxyvitamin D levels in children with SCD | 3 months follow up
  Serum levels of 25 Hydroxyvitamin D
Frequency of blood transfusion among children supplemented with vitamin D versus Placebo in children with sickle cell anaemia | 3 months follow up
  The number of children requiring blood transfusion during follow up and the episodes per child

SECONDARY OUTCOMES:
Incidence of vaso-occlusive crises (VOC) | 3 months follow up
  Incidence of painful vaso-occlusive crises
Incidence of acute severe respiratory illnesses | 3 months follow up
  Incidence of cough associated with difficult breathing confirmed as pneumonia or acute chest syndrome by a health worker
Severe adverse events | 3 months follow up
  Serious adverse events for example severe diarrhoea and vomiting with dehydration.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Ndeezi, PhD, Principal Investigator — Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant information may be shared with other researchers.
Supporting Information: CSR
Time Frame: within one year and the sharing period could extend beyond this period
Access Criteria: If requested by other researchers who have carried out similar studies for a meta-analysis

REFERENCES:
- [Background] Hyacinth HI, Gee BE, Hibbert JM. The Role of Nutrition in Sickle Cell Disease. Nutr Metab Insights. 2010 Jan 1;3:57-67. doi: 10.4137/NMI.S5048. PMID 21537370
- [Background] Nolan VG, Nottage KA, Cole EW, Hankins JS, Gurney JG. Prevalence of vitamin D deficiency in sickle cell disease: a systematic review. PLoS One. 2015 Mar 3;10(3):e0119908. doi: 10.1371/journal.pone.0119908. eCollection 2015. PMID 25734582
- [Background] Dougherty KA, Schall JI, Bertolaso C, Smith-Whitley K, Stallings VA. Vitamin D Supplementation Improves Health-Related Quality of Life and Physical Performance in Children with Sickle Cell Disease and in Healthy Children. J Pediatr Health Care. 2020 Sep-Oct;34(5):424-434. doi: 10.1016/j.pedhc.2020.04.007. Epub 2020 Jun 5. PMID 32507538
- [Result] Ndeezi G, Kiyaga C, Hernandez AG, Munube D, Howard TA, Ssewanyana I, Nsungwa J, Kiguli S, Ndugwa CM, Ware RE, Aceng JR. Burden of sickle cell trait and disease in the Uganda Sickle Surveillance Study (US3): a cross-sectional study. Lancet Glob Health. 2016 Mar;4(3):e195-200. doi: 10.1016/S2214-109X(15)00288-0. Epub 2016 Jan 29. PMID 26833239